CLINICAL TRIAL: NCT00142155
Title: Correlation of Fc Gamma RIIIA Receptor Expression and Response to Rituximab and Other Monoclonal Antibodies in Patients With Waldenstrom's Macroglobulinemia
Brief Title: Correlation of FC Gamma RIIIA Receptor Response in Patients With Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Other Study IDs: 02-075
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: monoclonal antibody; Fc gamma RIII receptor expression; rituximab
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Rituximab; Antibodies, Monoclonal

INTERVENTIONS:
Drug: Rituximab
Drug: monoclonal antibodies

SUMMARY:
The purpose of this study is to determine if the type of Fc gamma RIIIa receptor that a particular patient's immune cells possess influences how they respond to rituximab and other monoclonal antibodies.

DETAILED DESCRIPTION:
* A medical data collection survey sheet will be filled out by the patient or doctor with medical information pertaining to how the patient responded to rituximab and other monoclonal antibodies for use in this study.
* Blood work will be performed to analyze the blood by molecular technology to find the kind of Fc gamna RIIIa receptor the patient possess and correlate these findings with the outcome of treatment with rituximab or other monoclonal antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with rituximab or other monoclonal antibodies for Waldenstrom's macroglobulinemia

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2002-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Treon, MD, MA, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States